CLINICAL TRIAL: NCT06660537
Title: Effects of Balloon-blowing Exercises in 90/90 Bridge Position With a Ball on Pulmonary Function Among Asthmatic Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/37
Record Dates: First submitted 2024-10-24; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-09

CONDITIONS: Asthma
Keywords: Dyspnea, asthma, spirometry, quality of life, oxygen saturation
MeSH Terms: conditions — Asthma; Dyspnea

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial having two groups. One group will receive (interventional group) balloon-blowing exercises in 90/90 bridge position with a ball and the other group (control group) will receive buteyko breathing exercises.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): In this group patients will undergo balloon-blowing exercises in the 90/90 bridge position with a ball. In this intervention, patients lie on back with feet against a wall and knee bent at 90 degrees, holding a ball between their knees. While extending one arm overhead and holding a balloon in the other hand, perform a pelvic tilt without lifting their backoff the mat. Inhale through the nose, exhale into the balloon for four breaths, then remove the balloon and repeat the sequence four times. The 4-week protocol includes three supervised sessions per week, each supervised by a physiotherapist. Progress will be monitored regularly to evaluate improvements throughout the intervention.
  Interventions: Procedure: Balloon-blowing exercises in 90/90 bridge position with a ball.
- Control group (Experimental): In this group, patient will receive Buteyko breathing exercises consists of two main exercises; the control pause and the maximum pause .For control pause, patient exhale, plug the nose, and hold their breath until they feel the urge to breathe, then inhale and breathe normally for 10 seconds.In Maximum pause, patient exhale,plug their nose ,and hold their breath as long as posiible, aiming for double the control pause time, then inhale and breath normally for 10 seconds.This is a 4-week protocol with three sessions per week.Pre- and post- intervention values will be recorded to assess progress.n.
  Interventions: Procedure: Buteyko breathing exercises management

INTERVENTIONS:
Procedure: Balloon-blowing exercises in 90/90 bridge position with a ball. — In this group patients will undergo balloon-blowing exercises in the 90/90 bridge position with a ball. In this intervention, patients lie on back with feet against a wall and knee bent at 90 degrees, holding a ball between their knees. While extending one arm overhead and holding a balloon in the other hand, perform a pelvic tilt without lifting their back off the mat. Inhale through the nose, exhale into the balloon for four breaths, then remove the balloon and repeat the sequence four times. The 4-week protocol includes three supervised sessions per week, each supervised by a physiotherapist. Progress will be monitored regularly to evaluate improvements throughout the intervention.
  Arms: Interventional group
Procedure: Buteyko breathing exercises management — In this group, patients will receive Buteyko breathing exercises, which consist of two main exercises; the control pause and the maximum pause. For control pause, patients exhale, plug the nose, and hold their breath until they feel the urge to breathe, then inhale and breathe normally for 10 seconds. In Maximum pause, patients exhale, plug their nose, and hold their breath as long as possible, aiming for double the control pause time, then inhale and breath normally for 10 seconds. This is a 4-week protocol with three sessions per week. Pre- and post-intervention values will be recorded to assess progress.
  Arms: Control group

SUMMARY:
In asthma, the airways in the respiratory system can experience inflammation and constriction, causing increased difficulty in expelling air during exhalation. This results in disruptions to respiratory parameters, exercise intolerance, and a diminished overall quality of life.Engaging in balloon-blowing exercises while in a 90/90 bridge position with the use of a ball will lead to enhanced pulmonary function and quality of life in individuals with asthma.

DETAILED DESCRIPTION:
Asthma attacks and labored breathing can cause strain and weakness in the diaphragm, the main muscle supporting breathing, as well as the muscles of core.

The study objective is to determine the effects of balloon-blowing exercises in 90/90 bridge posotion with a ball on pulmonary function and quality of life among asthmatic patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults: aged (18-59 years)
* Gender: Both male and females
* Grade1- Grade 4 on Modified MRC dyspnea scale
* Asthma severity ( level 1 mild intermediate, levell 2 mild persistent)

Exclusion criteria:

* Level 3 and above asthmatics or status asthmatics.
* Any congenital deformities of chest wall/ Heart/ Lungs.
* Demonstrated neuromuscular or neurological deficit/ chest wall deformity.
* Cardiopulmonary diseases including coronary artery disease(CAD), Pulmonary HTN, ------Aortic Stenosis, regurgitation, etc.
* Any Autoimmune disease with manifestations of Chest wall/ heart/ Lungs.
* Any recent cardiothoracic or abdominal surgery or sternotomy.
* Recent history of the blunt chest wall or abdominal trauma.
* Unstable hemodynamic parameters (arterial pressure >140mmhg systolic and >90mmhg for diastolic).
* Pregnancy

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
pulmonary function test | 4 weeks
  Evaluation will be done using Spirometry
Dyspnea | 4 weeks
  Evaluation will be done using mMRC scale
Quality of life of patient | 4 Weeks
  Quality of life will be evaluated by asthma quality of life questionnaire with standardized Activities AQLQ(S)
Oxygen Saturation | 4 Weeks
  Oxygen saturation will be evaluated by pulse oximeter

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan